CLINICAL TRIAL: NCT02224209
Title: Comparison of Staged Angioplasty v.s. Routine Single-stage Stenting (CAS) in the Treatment of Patients With Carotid Artery Stenosis at High Risk of Hyperperfusion (STEP）: A Randomized Controlled Trial
Brief Title: Comparison of Staged Angioplasty and Routine Single-stage Stenting (CAS) in the Treatment of Carotid Artery Stenosis
Acronym: STEP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Zhongrong Miao, Director of Department of Intervention, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTH-STEP
Record Dates: First submitted 2014-08-08; First posted 2014-08-25 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Carotid Artery Stenosis
Keywords: Carotid artery stenosis; High risk of hyperperfusion; Staged angioplasty; Routine single-stage stenting
MeSH Terms: conditions — Carotid Stenosis | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Staged angioplasty (Experimental): Using Abbott EPD systems (Accunet/Emboshield), a balloon, stent
  Method of stage-1 angioplasty
  The stent can be placed into the distal stenosis under Abbott EPD systems (Accunet/Emboshield) if distal filter cannot be used, balloon angioplasty can be performed under proximal protection device; Use a balloon with diameter of 2mm × 2cm for stage-1 dilation until angiography shows residual stenosis <70%.
  Method of stage-2:
  The stent systems (Acculink/Xact) can be placed into the distal stenosis under Abbott EPD systems (Accunet/Emboshield); Use an Abbott balloon (diameter of 4 ~ 6mm) for pre-dilation or post-dilation; After the placement of stent, the angioplasty is a success when residual stenosis is <30%.
  Interventions: Device: Abbott EPD systems (Accunet/Emboshield), a balloon, stent
- Routine single-stage CAS (Active Comparator): Using a balloon, stent
  Routine stenting procedure:
  The stent systems (Acculink/Xact) can be placed into the distal stenosis under Abbott EPD systems (Accunet/Emboshield); Use an Abbott balloon (diameter of 4 ~ 6mm) for pre-dilation or post-dilation; After the placement of stent, the angioplasty is a success when residual stenosis is <30%.
  Interventions: Device: a balloon, stent

INTERVENTIONS:
Device: Abbott EPD systems (Accunet/Emboshield), a balloon, stent — Standard method of endovascular interventional treatment:
  Method of stage-1 angioplasty
  1. The stent can be placed into the distal stenosis under Abbott EPD systems (Accunet/Emboshield) if distal filter cannot be used, balloon angioplasty can be performed under proximal protection device;
  2. Use a balloon with diameter of 2mm × 2cm for stage-1 dilation until angiography shows residual stenosis <70%.
  Method of stage-2:
  1. The stent systems (Acculink/Xact) can be placed into the distal stenosis under Abbott EPD systems (Accunet/Emboshield);
  2. Use an Abbott balloon (diameter of 4 ~ 6mm) for pre-dilation or post-dilation;
  3. After the placement of stent, the angioplasty is a success when residual stenosis is <30%.
  Other Names: Abbott Stent System
  Arms: Staged angioplasty
Device: a balloon, stent — Routine stenting procedure:
  1. The stent systems (Acculink/Xact) can be placed into the distal stenosis under Abbott EPD systems (Accunet/Emboshield);
  2. Use an Abbott balloon (diameter of 4 ~ 6mm) for pre-dilation or post-dilation;
  3. After the placement of stent, the angioplasty is a success when residual stenosis is <30%.
  Other Names: Abbott Stent System
  Arms: Routine single-stage CAS

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of staged carotid angioplasty v.s. routine single-stage carotid artery stenting in Chinese patients with carotid artery stenosis at high hyperperfusion risk in peri-procedural period.

DETAILED DESCRIPTION:
1. Data Quality

   Before the initiation of the study sites, Cerebrovascular Disease Center of Beijing Tiantan Hospital will verify whether the investigators are qualified, inspect the study site's facilities, and inform the investigators of their responsibilities, as well as how to correctly and completely fill related documents. Through investigator training sessions, the investigators and their teams will understand the trial protocol, CRF and trial process, etc. Then start-up visit at each site will be initiated.

   Trial monitors will pay start-up visit to the site, and pay the first inspection visit as soon as possible after the screening/randomization of the first patient. Afterwards, the monitors will pay inspection visits regularly until the trial visits end. They need to directly refer to source data to verify the accurate of CRF filling and conduct inspection/audits.

   Data entered into the CRF shall be subject to examination of internal consistency (within known classification and scope), external inspection (data are consistent with the patient's other known data) and trend consistency (data changes do not exceed the allowable range. For example, excess weight loss prompts changes in dietary status). The contents of trial database include data collected by each site, abnormal data and delayed data in progress tracking.
2. File Data

   Data entered into the CRF must be able to be verified by source data, or directly entered into the CRF. In this case, the data in the CRF can be regarded as source data, and used for subsequent data confirmation. Required data of all patients' continued treatment shall also be routinely recorded in their medical records. The site's investigators shall clearly make patients' medical records that the patient is participating in a clinical trial, and also require any other medical staff for treatment of the patient to contact the trial contact persons before treatment. To this end, the investigators shall provide their contact information. If a patient preserves his/her medical records on his/her own, the study site shall preserve a copy of all trial-related data. Unless related data or information is directly recorded in the CRF, all research data must be recorded in patients' medical records (or research documents), and entered into the CRF as early as possible. Source data to be verified and primary documents used for such purpose must be preserved. Patients' research documents and all source data shall be preserved until a notice for destruction is received from the sponsor.
3. Statistical Method and Sample Size

   3.1 Statistical Analysis

   This study is powered on the primary endpoint of hyperperfusion syndrome (HPS) rate at 30 days post CAS procedure. Superiority analysis will be performed using a two-sample t-test at a two-sided 5% alpha level. All secondary endpoints will be descriptively compared between the two treatment arms.

   All analyses will be performed on the Per-Protocol (PP) population. The PP population will consist of patients who have received the treatment per randomization without major protocol deviations.

   X2 test is adopted for statistical analysis of two groups of results, supplemented by compliance with the protocol and actual treatment analysis. The following confounding factors will be considered in the analysis to determine the effect of different preset confounding factors on prognosis:
   * Age;
   * Sex;
   * Blood pressure;
   * Degree, location, diameter and length of lesion stenosis;
   * Cerebrovascular collateral compensatory conditions;
   * Cerebral hemodynamics of the culprit side;
   * Cerebrovascular reserve or cerebrovascular autoregulation status of the culprit side;
   * Diameter and pressure of balloon for stage-1 balloon angioplasty;
   * Carotid angioplasty experience of the operating site or doctor.

   Appropriate methods will be employed to summarize and analyze patients' baseline characteristics, safety and other indicators during the trial (including treatment interruption/termination, lifestyle assessment, concomitant medication, etc.). Multi-variant method is employed to analyze the effect of demographics and other factors on primary results. All details of statistical analysis are shown in the separate 'Statistical Analysis Plan'(SAP).

   3.2 Sample Size

   The sample size calculation for the primary endpoint of HPS rate 30 days post CAS procedure is based on the following assumptions:

   Two-tailed superiority test a = 0.05 Power = 90% Randomization ratio is 1 (staged angioplasty arm): 1 (routine single-stage CAS arm) The rate of HPS rate was expected to be 0.16 per subject during the procedure in the regular CAS arm for high hyperperfusion risk patients based on previous studies.

   The rate of HPS rate was presume to be 0.02 per subject during the procedure in the staged CAS arm for high hyperperfusion risk patients depended on the study by Yoshimura, Kyung Mi Lee and us.

   A total of 150 subjects were estimated to be required. Given the above assumptions, a sample size of 150 (75 Staged CAS: 75 regular CAS) will be required. To account for an estimated 5% dropout rate, approximately 158 patients will be enrolled. Of these 158 patients, 79 will be randomized to the Staged CAS arm and 79 will be randomized to the regular CAS arm.

   The sample size calculation was performed using SAS software, version 9.3 (SAS Institute).
4. Collection of data during the procedure

   * Nerve function evaluation
   * NIHSS
   * mRS
   * Blood pressure
   * TCD
   * Laboratory examination
   * CT, MR

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 40~80 years of age
* Patient with symptomatic carotid stenosis (defined as stroke/TIA of the patient within 90 days while he/she is taking at least one antithrombotic drug or under other intervention on vascular risk factors like hypertension or hyperlipidemia)
* DSA shows percent carotid stenosis≥90% (quantification of the stenosis according to NASCET method); or near occlusion
* Angiogram shows insufficient collateral circulation in the culprit vessel surrounding area:

  1. Cerebral CT perfusion imaging shows hypo-perfusion of the culprit vessel surrounding area, and
  2. DSA shows collateral circulation assessment < 2, and
  3. MRI cerebral imaging shows hemodynamic ischemic lesion
* CT perfusion imaging shows cerebral blood flow of the culprit side is of 20% lower than the other lateral brain
* Lesion length at the narrowest part < 25mm

Note: Grading of angiographic collateral circulation

* Grade 0: No collateral circulation in the area dominated by the culprit vessel
* Grade 1: Slow collateral circulation in the surrounding areas, but filling defects exist
* Grade 2: Fast collateral circulation, but some areas still have filling defects
* Grade 3: Collateral circulation is slow, but complete filling can be seen in the vein at a late stage
* Grade 4: Complete and fast collateral circulation, without any filling defect

Exclusion Criteria:

* Diffusive stenosis of the cerebral artery
* MRI cerebral imaging shows perforating artery occlusion
* Cerebral hemorrhage at the culprit vessel surrounding area within 6 weeks; potential thrombus from the heart
* Subsequent cerebral tumor, cerebral aneurysm, or arteriovenous abnormality
* Known contraindication to heparin, aspirin, ticlopidine, a aesthetic, and contrast; blood hemoglobin < 10g/dl, blood platelet < 100000
* Severe nerve dysfunction in the culprit vessel surrounding area after a cerebral infarction (mRS≥3)
* INR > 1.5 (irreversible), uncorrectable bleeding risk factors, life expectancy < 1 year
* Women in pregnant or breast feeding
* Committee adjudicating the inclusion criteria finds the patient is unsuitable for the staged angioplasty for carotid artery stenosis
* Unsuccessful placement of proximal or distal EPD during the procedure
* The target vessel angle≧45
* Participate in other clinical trials within three months

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-10 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Cerebral hyperperfusion syndrome or cerebral hemorrhage | Within 30 days after CAS procedure or after stage-1 balloon angioplasty procedure and after stage-2 CAS procedure.
  * Staged angioplasty arm: cerebral hyperperfusion syndrome or cerebral hemorrhage within 30 days after stage-1 balloon angioplasty procedure and after stage-2 CAS procedure.
  * Regular single-stage CAS arm: cerebral hyperperfusion syndrome or cerebral hemorrhage within 30 days after CAS procedure

SECONDARY OUTCOMES:
Cerebral hyperperfusion syndrome or cerebral hemorrhage attributed to the target vessel within 30 days after stage-1 balloon angioplasty or stage-2 CAS procedure. | within 30 days after stage-1 balloon angioplasty or stage-2 CAS procedure
Acute success of the culprit vessel after stage-1 balloon angioplasty (Diameter stenosis < 70%). | one year
Cerebral hyperperfusion syndrome attributed to non-culprit vessels within 30 days to 1 year post procedure. | one year
Any intracerebral hemorrhage, subarachnoid hemorrhage, or intraventricular hemorrhage within 30 days to 1 year post procedure. | one year
Myocardial infarchtion (MI) | one year
Major non-stroke hemorrhage (eg. Epidural hemorrhage, intradural hemorrhage, or other major systemic bleedings) | one year
Death at 30 days post procedure | one year
Stoke resulting in deformity | one year
Any stroke or death | one year

CONTACTS AND LOCATIONS:
Overall Officials: Zhongrong Miao, M.D., Study Director — Beijing Tian Tan Hospital, Capital Medical University; Yongjun Wang, M.D., Study Director — Beijing Tian Tan Hospital
Locations (1):
- Beijing Tian Tan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Mo D, Jia B, Shi H, Sun Y, Liu Q, Fan C, Deng J, Yuan J, Wu W, Jiang C, Zhang G, Du H, Ma N, Gao F, Sun X, Song L, Liu L, Peng G, Wang Y, Wang Y, Miao Z; STEP Study Group. Staged angioplasty versus regular carotid artery stenting in patients with carotid artery stenosis at high risk of hyperperfusion: a randomised clinical trial. Stroke Vasc Neurol. 2021 Mar;6(1):95-102. doi: 10.1136/svn-2020-000391. Epub 2020 Sep 24. PMID 32973113